CLINICAL TRIAL: NCT04176003
Title: OMERACT Core Domain Set Selection for Calcium Pyrophosphate Deposition (CPPD): Exploring Patient and Stakeholder Perspectives on Outcome Domains
Brief Title: Perspectives on CPPD Outcome Domains
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 19061
Record Dates: First submitted 2019-10-17; First posted 2019-11-25 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: CPPD - Calcium Pyrophosphate Deposition Disease
Keywords: Calcium Pyrophosphate Deposition Disease; Outcome measures; Qualitative research
MeSH Terms: conditions — Chondrocalcinosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with CPPD
  Interventions: Other: Qualitative interview; Other: Member checking
- Healthcare professionals working with CPPD patients
  Interventions: Other: Qualitative interview; Other: Member checking
- Stakeholders working on behalf of CPPD patients
  Interventions: Other: Qualitative interview; Other: Member checking

INTERVENTIONS:
Other: Qualitative interview — Qualitative interview to explore experiences and perceptions of living with CPPD, and outcome measures to use in future studies
Other: Member checking — Participants will be sent a short report with the researchers' findings from the qualitative interview, and asked to check the accuracy of these and provide brief written feedback.

SUMMARY:
The purpose of this study is to obtain patient and stakeholder perspectives on what outcome measures should be included in future trials on CPPD (Calcium PyroPhosphate Deposition), a common form of inflammatory arthritis. This will form part of a wider OMERACT (Outcome Measures in Rheumatology) study, involving multiple international sites, to determine a core domain set (an agreed set of outcome measures) for this disease.

In the UK, up to 10 patients with CPPD and their caregivers, healthcare professionals who care for patients with CPPD, and other stakeholders, which may include government organisations, non-government organisations, pharmaceutical representatives and health advocacy groups, will be invited to participate in a single, semi-structured interview.

Interviews will be face-to-face or telephone, last up to one hour and digitally audio-recorded. For patients and their caregivers, interviews will explore their lived experience of CPPD, its impact on their daily lives, and the perceived relevance of outcome measures used in previous studies. For healthcare professionals and other stakeholders, interviews will explore their experience dealing with patients with CPPD, how they perceive CPPD impacts patient lives, and the perceived relevance of the outcome measures used in previous studies.

Following analysis of the data, participants will be sent a short report with the researchers' findings, and asked to check the accuracy of these and provide brief written feedback.

Interviews will also take place with patients, caregivers, healthcare practitioners and stakeholders at the other international sites where ethics committee approval will be sought locally. It is anticipated that around 30 participants will be recruited across all sites. Analysis of all interviews will be primarily conducted and managed at the UK site.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* People with a diagnosis of CPPD of any form and/or their caregiver (includes acute CPP crystal arthritis (pseudogout), chronic CPP crystal arthritis, crowned dens syndrome, and osteoarthritis with CPPD)
* Ability to give informed consent
* Age over 18 years

Healthcare professionals:

* A healthcare professional (nurse, GP or hospital doctor) who cares or has cared for patients with CPPD

Other stakeholders:

* Government organisations, non-government organisations, pharmaceutical representatives and health advocacy groups

Exclusion Criteria:

* Dementia
* Terminal illness
* Unable to give informed consent
* Stroke with receptive or expressive dysphasia
* Severe enduring mental illness
* Autoimmune rheumatic disease such as rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, gout
* Total joint replacement in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CPPD, healthcare practitioners who work with patients with CPPD, and stakeholders who work on behalf of those with CPPD
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Patient and stakeholders perception of core outcome domains identified from a systematic literature review of clinical studies of patients with CPPD | 1 day
  This is a qualitative interview study, the primary aim is to collect patient and stakeholder perspectives on existing outcome measures of CPPD. Currently there are no recommended core outcome measure sets for CPPD and this work is being undertaken within the framework of OMERACT. Thematic analysis will be undertaken of interview transcripts and therefore there is no defined outcome measure.

SECONDARY OUTCOMES:
Experience of living with and perceptions of CPPD, and perceived impact of symptoms on daily life | 1 day
  This is a qualitative interview study, the secondary aim is to collect patients' experiences of living with CPPD as well as their and stakeholders perception of the impact of CPPD symptoms, to identify any further outcome measures that could be used in studies of CPPD. Currently there are no recommended core outcome measure sets for CPPD and this work is being undertaken within the framework of OMERACT. Thematic analysis will be undertaken of interview transcripts and therefore there is no defined outcome measure. There is no specific recall period for which experiences will be assessed as this will be dependent on each individual's disease duration.

CONTACTS AND LOCATIONS:
Overall Officials: A Abhishek, Principal Investigator — University of Nottingham
Locations (1):
- Academic Rheumatology, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided